CLINICAL TRIAL: NCT05863741
Title: Does Personalized Soft Tissue Balance Data Improve Outcomes in Patients Undergoing Medially Stabilized Knee Arthroplasty? A Prospective, Randomized Study Investigating the Clinical Utility of the NextAR Navigation System (NextAR).
Brief Title: Clinical Utility and Gait Analysis of NextAR System AUS
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P02.022.01
Record Dates: First submitted 2023-04-26; First posted 2023-05-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control study: patients will be operated with conventional instrumentation
  Interventions: Device: Implantation of GMK Sphere with conventional instrumentation
- NextAR study: patients will be operated using the NextAR guidance system
  Interventions: Device: Implantation of GMK Sphere using the NextAR guidance system

INTERVENTIONS:
Device: Implantation of GMK Sphere with conventional instrumentation — Implantation of GMK Sphere with conventional instrumentation (control group)
  Groups: control study
Device: Implantation of GMK Sphere using the NextAR guidance system — Implantation of GMK Sphere using the NextAR guidance system (NextAR group)
  Groups: NextAR study

SUMMARY:
This study titled "Does Personalised Soft Tissue Balance Data Improve Outcomes in Patients Undergoing Medially Stabilised Arthroplasty? A Prospective, Randomised Study Investigating the Clinical Utility of the NextAR navigation system (NextAR)" is a randomised, single blinded, prospective cohort study with the primary aim determine the clinical utility of the NextAR system data in providing soft tissue balance patterns to enable prosthesis implants to resemble more native knee alignment.

DETAILED DESCRIPTION:
This study titled "Does Personalised Soft Tissue Balance Data Improve Outcomes in Patients Undergoing Medially Stabilised Arthroplasty? A Prospective, Randomised Study Investigating the Clinical Utility of the NextAR navigation system (NextAR)" is a randomised, single blinded, prospective cohort study with the primary aim determine the clinical utility of the NextAR system data in providing soft tissue balance patterns to enable prosthesis implants to resemble more native knee alignment.

The aims of this study are:

* To determine the clinical utility of the NextAR system data in providing soft tissue balance patterns to enable prosthesis implants to resemble more native knee alignment
* To determine whether NextAR system data contributes to improving patient outcomes and knee kinematics following TKR surgery, by providing greater flexion range that is equivalent to native knee motion.
* To assess clinical outcomes measured by standardised assessments, including radiographic evidence, the Forgotten Joint Score (FJS), the Oxford Knee Score (OKS), International Knee Documentation Committee (IKDC) and European Quality of Life Five Dimensions - Five Levels (EQ5D-5L) questionnaires.
* Determining the kinematics of the replaced knee as measured by 3D gait analysis.

According to study protocol, clinical evaluation is performed preoperatively and postoperatively at 6 weeks, 6 months, 1, and 2 years with the use of the Forgotten Joint Score (FJS), Oxford Knee Score (OKS), International Knee Documentation Committee (IKDC) and European Quality of Life Five Dimensions - Five Levels (EQ5D-5L).

CT scan is performed preoperatively and at 6-weeks after surgery, while X-ray assessment is performed at baseline and at the 1-year follow up.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee suitable for total knee arthroplasty.
* Aged over 18 years.

Exclusion Criteria:

* Unsuitable for TKR due to chronic infection, medical disease, inability to consent, inability to attend for post-operative follow-up, significant psychiatric issues, substance abuse issues
* Previous reconstructive/fracture/arthroplasty surgery on affected knee
* Active inflammation arthropathy
* Significant extra articular deformity
* Morbidly Obese (BMI >40)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The trial will include two groups of 50 patients in each group. This is based on a power calculation assuming a difference in Forgotten Join Score of greater than 5 points. This calculation allows for a loss to follow-up of 10%. The study will conclude once the patients involved have completed 2 years of follow-up.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Determine whether NextAR system data contributes to change patient outcomes using the Forgotten Joint Score | pre-op, 6 weeks, 6 months, 1 year, 2 years
  To determine whether NextAR system data contributes to change patient outcomes using the Forgotten Joint Score
  - Forgotten Joint Score measures the patient's ability to forget about the joint as a result of successful treatment and is based on the premise that the best arthroplasty is one the patient forgets. This score goes from a minimum of 0 to a maximum of 100 points.

SECONDARY OUTCOMES:
To determine whether NextAR system data contributes to change patient outcomes using the EQ5D-5L | pre-op, 6 weeks, 6 months, 1 year, 2 years
  To determine whether NextAR system data contributes to change patient outcomes using the EQ5D-5L
  The EQ5D-5L comprises of 6 questions survey that measures generic health-related quality of life. This score goes from a minimum of 0 to a maximum of 1 points.
Determining the kinematics of the replaced knee as measured by 3D gait analysis. | pre-op, 1 year
  The purpose of the gait analysis will be to assess the variation in kinematics between the patients replaced knee (in both study groups) compared to normal knee kinematic data reported in the literature. The hypothesis being tested is that alteration of component position to give more normal ligament tension, will more resemble normal knee kinematics. (n=20) will be sufficient to conduct the gait analysis. These patients will be selected from the overall cohort for enrolment at 12 months post-surgery and matched for age, gender, BMI and osteoarthritis pattern. The comparison will involve comparing the average kinematic data values obtained in group 1 (NextAR data provided at surgery) vs the reported values in the literature and the same analysis will be repeated for patients in group 2 (NextAR data not provided at surgery).comparison will be made between the two groups in terms of which more closely replicates the kinematics of the non-arthritic knee
To determine whether NextAR system data contributes to change patient outcomes using the Oxford Knee Score | pre-op, 6 weeks, 6 months, 1 year, 2 years
  To determine whether NextAR system data contributes to change patient outcomes using the Oxford Knee Score
  the Oxford Knee Score is a questionnaire that has been specifically developed to assess knee function and pain. It is short, reproducible and extensively referenced in orthopaedic literature, making it a preferred tool for studies. This score goes from a minimum of 0 to a maximum of 48 points.
To determine whether NextAR system data contributes to change patient outcomes using the Forgotten Joint Score using the International Knee Documentation Committee | pre-op, 6 weeks, 6 months, 1 year, 2 years
  To determine whether NextAR system data contributes to change patient outcomes using the Forgotten Joint Score using the International Knee Documentation Committee
  International Knee Documentation Committee is questionnaire that evaluates physical activity, level of pain and knee functionality in sporting activities. This score goes from a minimum of 0 to a maximum of 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Jeffcote, Principal Investigator — Fremantle Hospital
Locations (1):
- Fremantle Hospital, Fremantle, Australia

IPD SHARING:
Plan to Share IPD: No